CLINICAL TRIAL: NCT04597021
Title: Performing Central Venous Catheters in Neonates and Small Infants Undergoing Cardiac Surgery Using a Wireless Transducer for Ultrasound Guidance: a Prospective, Observational Pilot Study
Brief Title: Wireless US-guided CVC Placement in Infants
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Judith Schiefer, MD; PhD., Medical University of Vienna
Other Study IDs: 1386/2018
Record Dates: First submitted 2020-10-15; First posted 2020-10-22 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Wireless Ultrasound; Central Venous Catheter; Congenital Heart Disease in Children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: use of a wiresless US transducer — to (evaluate the practicability of applying a wireless US transducer for central venous catheter-placement in these patients.

SUMMARY:
Background: Neonates and small infants with congenital cardiac disease undergoing cardiac surgery represent major challenges facing pediatric anesthesia and perioperative medicine. Aims: We here aimed to investigate the success rates in performing ultrasound guided central venous catheter insertion (CVC) in neonates and small infants undergoing cardiac surgery, and to evaluate the practicability and feasibility of thereby using a novel wireless ultrasound transducer (WUST).

Methods: Thirty neonates and small infants with a maximum body weight of 10 kg and need for CVC before cardiac surgery were included in this observational trial and were subdivided into two groups according to their weight: < 5 kg and ≥5 kg. Cannulation success, failure rate, essential procedure related time periods, and complications were recorded and the clinical utility of the WUST was assessed by a 5-point Likert scale.

ELIGIBILITY:
Inclusion Criteria:

neonates and small infants with a maximum body weight of 10 kg and need for insertion of a CVC before cardiac surgery at our institution

Exclusion Criteria:

* missing consent for study participation >10 kg body weight
* emergency surgery
* central venous catheter in situ

Max Age: 2 Years | Sex: All
Age Groups: Child
Study Population: neonates and small infants with a maximum body weight of 10 kg and need for insertion of a CVC before cardiac surgery at our institution
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Rate of success using a wireless US for pediatric CVC | during cardiac surgery
  Clinical applicability of a wireless US transducer for CVC insertion for pediatric cardiac surgery

CONTACTS AND LOCATIONS:
Overall Officials: Judith Schiefer, MD, Ph, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schiefer J, Lichtenegger P, Zimpfer D, Hutschala D, Kuessel L, Felli A, Hornykewycz S, Faybik P, Base E. Performing central venous catheters in neonates and small infants undergoing cardiac surgery using a wireless transducer for ultrasound guidance: a prospective, observational pilot study. BMC Pediatr. 2021 Aug 13;21(1):341. doi: 10.1186/s12887-021-02822-w. PMID 34389009